CLINICAL TRIAL: NCT01423084
Title: A Phase 3, Randomized, Comparative, Multicenter Observer-Blind Study Evaluating the Safety and Immunogenicity of Novartis Meningococcal B Vaccine Formulated With OMV Manufactured at Two Different Sites, in Healthy Adolescents Aged 11-17 Years
Brief Title: Safety and Immunogenicity of Novartis Meningococcal B Vaccine Formulated With OMV Manufactured at Two Different Sites, in Healthy Adolescents Aged 11-17 Years
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: V72_41
Record Dates: First submitted 2011-08-23; First posted 2011-08-25 (Estimated); Results first posted 2015-02-20 (Estimated); Last update posted 2015-02-20 (Estimated); Status verified 2015-02

CONDITIONS: Meningococcal Disease; Meningococcal Meningitis
Keywords: Meningococcal Meningitis; prevention, vaccination; adolescents
MeSH Terms: conditions — Meningococcal Infections; Meningitis, Meningococcal | interventions — 4CMenB vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MenB Lot 1 (Experimental): MenB vaccine Lot 1: 2 doses administered 1 month apart
  Interventions: Biological: Serogroup B meningococcal vaccine
- MenB Lot 2 (Active Comparator): MenB vaccine Lot 2: 2 doses administered 1 month apart
  Interventions: Biological: Serogroup B meningococcal vaccine

INTERVENTIONS:
Biological: Serogroup B meningococcal vaccine — All subjects will receive two rMenB+OMV NZ vaccinations one month apart and will be followed for a total of 2 months. Subjects will be randomized to 1 of 2 treatment arms to receive either two doses of rMenB+OMV NZ vaccine Lot 1 or two doses of rMenB+OMV NZ Lot 2.
  A total of 2 blood samples will be collected (at the first vaccination and 1 month after the 2nd vaccination). An additional blood draw will be collected in a subset of approximately 160 subjects (approximately 80 subjects in Group 1 and approximately 80 subjects in Group 2) at 2 weeks after the second vaccination

SUMMARY:
The primary objective of this study is to demonstrate the equivalence of rMenB+OMV NZ lot 1 to rMenB+OMV NZ lot 2 when administered to adolescents, as measured by human serum bactericidal activity (hSBA) geometric mean titers (GMTs) against 3 N. meningitidis serogroup B reference strains (H44/76, 5/99, and NZ98/254) and as measured by ELISA geometric mean concentrations (GMCs) against vaccine antigen 287-953, approximately 30 days after a primary vaccination course of two doses administered one month apart.

DETAILED DESCRIPTION:
Novartis will consider this study a success if, at one month following the second vaccination, the two-sided 95% CI of the ratio of the hSBA GMTs for each of 3 serogroup B reference strains (H44/76, 5/99, and NZ98/254) and the two-sided 95% CI of the ratio of the ELISA GMCs against vaccine antigen 287-953 are contained within the interval (0.5, 2.0).

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects (11-17 years of age inclusive) who have given their written assent and whose parents or legal guardians have given written informed consent at the time of enrollment
* who are available for all the visits scheduled in the study (i.e., not planning to leave the area before the end of the study period)
* in good health as determined by the outcome of medical history, physical examination and clinical judgment of the investigator.

Exclusion Criteria:

* History of any serogroup B meningococcal vaccination
* Current or previous, confirmed or suspected disease caused by N. meningitidis
* Exposure to an individual with any laboratory confirmed N. meningitidis infection within 60 days of enrollment
* Significant acute or chronic infection within the previous 7 days or fever (defined as axillary temperature ≥ 38.0 °C) within the previous day
* Antibiotic use within 3 days (72 hours) prior to enrollment
* Pregnancy or nursing (breastfeeding) mothers
* Females of childbearing age who have not used or do not plan to use acceptable birth control measures, for the 2 months duration of the study. If sexually active the subject must have been using one of the accepted birth control methods for at least 30 days prior to study entry
* Any serious chronic or progressive disease, Known or suspected impairment/alteration of the immune system
* Receipt of blood, blood products and/or plasma derivatives, or a parenteral immunoglobulin preparation within the previous 90 days
* History of severe allergic reactions after previous vaccinations or hypersensitivity to any vaccine component

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 344 (Actual)
Dates: Start 2011-08; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- Australia (6):
  - Royal Children's Hospital, Herston, Queensland
  - AusTrials Pty Ltd-Suites 6, 10 & 11, Peninsula Specialist Centre, Kippa-Ring, Queensland
  - AusTrials Pty Ltd-Suite 5, Level 1, 14 Primrose Street, Sherwood, Queensland
  - Women's and Children's Hospital, 72 King William Road, North Adelaide, South Australia
  - Murdoch Children's Research Institute-Level 5, 207 Bouverie St-University of Melbourne, Melbourne, Victoria
  - Telethon Institute for Child Heath Research-cnr, Hamilton Street and Roberts Road-Subiaco, Western Australia
- Canada (7):
  - TASC Research Services, 1-15243 91st Avenue, Surrey, British Columbia
  - Colchester Regional Hospital Colchester Research Group, 68 Robie Street, Truro, Nova Scotia
  - Albion Finch Medical Centre, 1620 Albion Road, Suite 106, Etobicoke, Ontario
  - Medicor Research Inc, 359 Riverside, Suite 200, Greater Sudbury, Ontario
  - SKDS Research Inc, 221-679 Davis Dr.Newmarket, Toronto, Ontario
  - Dr. Hartley Garfield Medicine Professional Corporation, 790 Bay Street, Suite 540, Toronto, Ontario
  - Devonshire Clinical Research INC, 423 Devonshire Ave., Suite 301, Woodstock, Ontario

REFERENCES:
- [Derived] Perrett KP, McVernon J, Richmond PC, Marshall H, Nissen M, August A, Percell S, Toneatto D, Nolan T. Immune responses to a recombinant, four-component, meningococcal serogroup B vaccine (4CMenB) in adolescents: a phase III, randomized, multicentre, lot-to-lot consistency study. Vaccine. 2015 Sep 22;33(39):5217-24. doi: 10.1016/j.vaccine.2015.06.103. Epub 2015 Jul 29. PMID 26232542

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Actual start date of recruiting was 30 August 2011. Subjects were recruited from 7 centres in Canada and 6 centres in Australia.
Pre-assignment Details: All subjects were enrolled in the trial.
Groups:
- 4CMenB_Rosia: Subjects received two doses of rMenB+OMV NZ vaccine from lot 1 manufactured at Rosia facility.
- 4CMenB_Siena: Subjects received two doses of rMenB+OMV NZ vaccine from lot 2 manufactured at Siena facility.
Period: Overall Study
Arm/Group | 4CMenB_Rosia | 4CMenB_Siena
Started | 170 | 174
Completed | 168 | 170
Not Completed | 2 | 4
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 2 | 3

BASELINE CHARACTERISTICS:
Population: adolescents aged 11-17 years
Groups:
- Total: Total of all reporting groups
Arm/Group | 4CMenB_Rosia | 4CMenB_Siena | Total
Number analyzed (Participants) | 170 | 174 | 344
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.6 (1.9) | 13.8 (1.8) | 13.7 (1.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 82 | 154
  Male | 98 | 92 | 190

OUTCOME MEASURES:

1. Primary Outcome: Human Serum Bactericidal Activity (hSBA) Geometric Mean Titers (GMTs) Against 3 Neisseria.Meningitidis (N. Meningitidis) Serogroup B Reference Strains.
Description: Consistency of the immune response of the two lots of rMenB+OMV NZ will be assessed at one month after the second vaccination based on the ratio of the vaccine lot hSBA GMTs for each of three serogroup B reference strains (H44/76, 5/99, and NZ98/254) and based on the ratio of Enzyme-linked Immunosorbent Assay (ELISA) GMCs for vaccine antigen 287-953. The equivalence interval will be (0.5, 2.0).
Time Frame: One month after the second vaccination (day 61)
Population: Per Protocol Set population
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 4CMenB_Rosia | 4CMenB_Siena
Number analyzed (Participants) | 147 | 151
Titers
  H44/76 strain | 111 [96 to 129] | 111 [96 to 128]
  NZ98/254 strain | 9.27 [7.44 to 12] | 11 [9.22 to 14]
  5/99 strain (N=152) | 183 [160 to 209] | 199 [174 to 227]
Statistical Analysis 1: Comparison: 4CMenB_Rosia vs 4CMenB_Siena; Equivalence of 2 different lots of rMenB+OMV NZ in terms of hSBA GMTs against H44/76 strain; Test type: Non-Inferiority or Equivalence — Two different lots of rMenB+OMV NZ are to be considered equivalent in terms of hSBA GMTs against H44/76 strain if the two sided 95% Confidence Interval (CI) between groups GMTs ratio at day 31 (ie, one month after the second vaccination) does not exceed the range 0.5 (lower limit) - 2.0 (higher limit); between groups ratio = 1, 95% CI 2-sided [0.82 to 1.23]
Statistical Analysis 2: Comparison: 4CMenB_Rosia vs 4CMenB_Siena; Equivalence of 2 different lots of rMenB+OMV NZ in terms of hSBA GMTs against 5/99 strain; Test type: Non-Inferiority or Equivalence — Two different lots of rMenB+OMV NZ are to be considered equivalent in terms of hSBA GMTs against 5/99 strain if the two sided 95% Confidence Interval (CI) between groups GMTs ratio at day 31 (ie, one month after the second vaccination ) does not exceed the range 0.5 (lower limit) - 2.0 (higher limit); between groups ratio = 0.92, 95% CI 2-sided [0.77 to 1.1]
Statistical Analysis 3: Comparison: 4CMenB_Rosia vs 4CMenB_Siena; Equivalence of 2 different lots of rMenB+OMV NZ in terms of hSBA GMTs against NZ98/254 strain; Test type: Non-Inferiority or Equivalence — Two different lots of rMenB+OMV NZ are to be considered equivalent in terms of hSBA GMTs against NZ 98/254 strain if the two sided 95% Confidence Interval (CI) between groups GMTs ratio at day 31 (ie, one month after the second vaccination ) does not exceed the range 0.5 (lower limit) - 2.0 (higher limit); between groups ratio = 0.81, 95% CI 2-sided [0.6 to 1.09]

2. Secondary Outcome: Percentage of Subjects in Each Lot With hSBA ≥ 1:5
Description: The percentage of subjects in each lot with hSBA ≥ 1:5 at one month after the second vaccination for each of the three reference strains (H44/76, 5/99, and NZ98/254) for each vaccine group
Time Frame: One month after the second vaccination (day 61)
Population: Per Protocol Set population
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | 4CMenB_Rosia | 4CMenB_Siena
Number analyzed (Participants) | 147 | 152
Percentage of subjects
  H44/76 strain (N=151) | 99 [96 to 100] | 99 [96 to 100]
  NZ98/254 strain (N=151) | 70 [62 to 77] | 79 [72 to 86]
  5/99 strain | 100 [98 to 100] | 100 [98 to 100]

3. Secondary Outcome: Geometric Mean Ratio (GMR) of GMTs Against Each of N. Meningitidis Serogroup B Reference Strains.
Description: The immune response of two different lots of rMenB+OMV NZ against each of N. meningitidis serogroup B test strains is evaluated in terms of GMR between GMTs (1month after the second vaccination vs baseline).
Time Frame: One month after the second vaccination (day 61)
Population: Per Protocol Set Population
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio of GMTs
Arm/Group | 4CMenB_Rosia | 4CMenB_Siena
Number analyzed (Participants) | 147 | 152
Ratio of GMTs
  H44/76 strain (N=151) | 104 [89 to 121] | 107 [92 to 124]
  NZ98/254 strain (N=151) | 8.63 [6.99 to 11] | 11 [8.99 to 14]
  5/99 | 156 [133 to 183] | 167 [143 to 195]

4. Secondary Outcome: Geometric Mean Ratio (GMR) of ELISA Geometric Mean Concentration (GMCs) Against Antigen 287-953
Description: The immune response of two different lots of rMenB+OMV NZ against antigen 287-953 is evaluated in terms of GMRs between ELISA GMCs (day 61 vs baseline).
Time Frame: One month after the second vaccination (day 61)
Population: Per Protocol Set Population
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio of GMTs
Arm/Group | 4CMenB_Rosia | 4CMenB_Siena
Number analyzed (Participants) | 145 | 152
Ratio of GMTs | 122 [103 to 143] | 153 [131 to 179]

5. Secondary Outcome: hSBA GMT Against 3 N. Meningitidis Serogroup B Reference Strains at Day 45.
Description: The immunogenicity of two different lots of rMenB+OMV NZ is evaluated in terms of hSBA GMT against 3 N. Meningitidis serogroup B reference strains at two weeks after last vaccination.
Time Frame: Two weeks after the second vaccination (day 45)
Population: Per Protocol Set, immunogenicity subset
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- MenB Lot 2: Subjects received two doses of rMenB+OMV NZ vaccine from lot 2 manufactured at Siena facility.
Arm/Group | 4CMenB_Rosia | MenB Lot 2
Number analyzed (Participants) | 76 | 71
Titers
  H44/76 strain | 187 [152 to 229] | 171 [139 to 210]
  NZ98/254 strain | 14 [10 to 18] | 20 [15 to 27]
  5/99 strain | 254 [206 to 314] | 339 [273 to 420]

6. Secondary Outcome: GMRs of GMT Against 3 N. Meningitidis Serogroup B Reference Strains at Day 45.
Description: The immunogenicity of two different lots of rMenB+OMV NZ is evaluated in terms of GMRs of GMT against 3 N.
  meningitidis serogroup B reference strains at two weeks after last vaccination.
Time Frame: Two weeks after the second vaccination (day 45)
Population: Per Protocol Set, Immunogenicity subset
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio of GMTs
Arm/Group | 4CMenB_Rosia | 4CMenB_Siena
Number analyzed (Participants) | 76 | 71
Ratio of GMTs
  H44/76 strain | 174 [138 to 219] | 157 [124 to 199]
  NZ98/254 | 13 [9.87 to 17] | 20 [15 to 26]
  5/99 strain | 214 [161 to 284] | 243 [183 to 325]

7. Secondary Outcome: Percentage of Subjects With hSBA ≥1:5 Against Each of N. Meningitidis Serogroup B Reference Strains at Day 45.
Description: The immune response of two different lots of rMenB+OMV NZ against each of N. Meningitidis serogroup B reference strains is evaluated in terms of percentages of subjects with hSBA ≥1:5 two weeks after the last vaccination.
Time Frame: Two weeks after the second vaccination (day 45)
Population: Per Protocol Population, immunogenicity subset
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | 4CMenB_Rosia | 4CMenB_Siena
Number analyzed (Participants) | 76 | 71
Percentage of subjects
  H44/76 strain | 100 [95 to 100] | 100 [95 to 100]
  NZ98/254 strain | 84 [74 to 92] | 96 [88 to 99]
  5/99 strain | 100 [95 to 100] | 100 [95 to 100]

8. Secondary Outcome: ELISA GMCs Against Vaccine Antigen 287-953 at Day 45.
Description: The immune response of two different lots of rMenB+OMV NZ is evaluated in terms of ELISA GMCs against vaccine antigen 287-953.
Time Frame: Two weeks after the second vaccination (day 45)
Population: Per Protocol Set, immunogenicity subset.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/ml
Arm/Group | 4CMenB_Rosia | 4CMenB_Siena
Number analyzed (Participants) | 76 | 71
IU/ml | 3742 [2994 to 4676] | 4798 [3825 to 6019]

9. Primary Outcome: ELISA Geometric Mean Concentration (GMCs) Against Vaccine Antigen 287-953
Description: as for outcome 8
Time Frame: One month after the second vaccination (day 61)
Population: Per Protocol Set population
Measure: Geometric Mean (95% Confidence Interval); unit: IU/ml
Arm/Group | 4CMenB_Rosia | 4CMenB_Siena
Number analyzed (Participants) | 147 | 152
IU/ml | 2729 [2338 to 3186] | 3291 [2829 to 3828]
Statistical Analysis 1: Comparison: 4CMenB_Rosia vs 4CMenB_Siena; Equivalence of 2 different lots of rMenB+OMV NZ in terms of hSBA GMTs; Test type: Non-Inferiority or Equivalence — Two different lots of rMenB+OMV NZ are to be considered equivalent in terms of ELISA GMCs against vaccine antigen 287-953 if the two sided 95% Confidence Interval (CI) between groups GMTs ratio at day 31 (ie, one month after the second vaccination ) does not exceed the range 0.5 (lower limit) - 2.0 (higher limit); between groups ratio = 0.83, 95% CI 2-sided [0.67 to 1.02]

10. Secondary Outcome: GMR of ELISA GMCs Against Antigen 287-953 at Day 45.
Description: The immune response of two different lots of rMenB+OMV NZ against antigen 287-953 is evaluated in terms of GMRs between ELISA GMCs (day 45 vs baseline).
Time Frame: Two weeks after the second vaccination (day 45)
Population: Per Protocol Set, immunogenicity subset
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio of GMTs
Arm/Group | 4CMenB_Rosia | 4CMenB_Siena
Number analyzed (Participants) | 74 | 71
Ratio of GMTs | 166 [130 to 213] | 217 [169 to 279]

11. Secondary Outcome: Number of Subjects Reporting Solicited Local and Systemic Adverse Events (AEs)
Description: Number of subjects reporting solicited local and systemic Adverse Events and other indicators of reactogenicity after any vaccination.
Time Frame: From day 1 to day 7 after any vaccination
Population: Safety Set
Measure: Number; unit: Number of subjects
Arm/Group | 4CMenB_Rosia | 4CMenB_Siena
Number analyzed (Participants) | 169 | 173
Number of subjects
  Any local | 163 | 170
  Induration | 65 | 75
  Pain | 162 | 170
  Erythema | 111 | 111
  Swelling | 80 | 74
  Any systemic | 136 | 150
  Nausea | 49 | 56
  Fatigue | 75 | 85
  Myalgia | 99 | 118
  Arthralgia | 28 | 44
  Headache | 75 | 89
  Fever (>= 38C) | 8 | 5
  Rash | 11 | 16
  Any other | 87 | 96
  Use of analgesics | 82 | 92

12. Secondary Outcome: Number of Subjects Reporting Unsolicited AEs
Description: Number of subjects reporting any Unsolicited AEs after any vaccination.
Time Frame: From day 1 to day 7 after any vaccination.
Population: Safety Set
Measure: Number; unit: Number of subjects
Arm/Group | 4CMenB_Rosia | 4CMenB_Siena
Number analyzed (Participants) | 169 | 173
Number of subjects | 56 | 55

13. Secondary Outcome: Number of Subjects Reporting SAEs and AE Leading to Withdrawal
Description: Number of subjects reporting any Serious AEs (SAEs), medically attended AEs and AEs that result in a subject's withdrawal from the study after any vaccination.
Time Frame: Throughout the study period.
Population: Safety Set
Measure: Number; unit: Number of subjects
Arm/Group | 4CMenB_Rosia | 4CMenB_Siena
Number analyzed (Participants) | 169 | 173
Number of subjects
  Serious Adverse Events | 0 | 0
  Adverse Events | 0 | 1

ADVERSE EVENTS:
Time Frame: SAEs were collected from day 1 through study termination, other AEs were collected from day 1 to day 7 after vaccination.
Arm/Group | 4CMenB_Rosia | 4CMenB_Siena
Serious Adverse Events (participants affected / at risk) | 0/169 | 0/173
Other Adverse Events (participants affected / at risk) | 165/169 | 171/173
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 4CMenB_Rosia (N=169) | 4CMenB_Siena (N=173)
injection site swelling (Investigations) | 80 (115) | 74 (107)
Headache (Nervous system disorders) | 75 (124) | 89 (159)
Fatigue (General disorders) | 75 (129) | 85 (138)
injection site induration (General disorders) | 65 (96) | 75 (107)
injection site erythema (General disorders) | 111 (177) | 111 (175)
injection site pain (General disorders) | 162 (337) | 170 (349)
nausea (Gastrointestinal disorders) | 49 (68) | 56 (77)
rash (Skin and subcutaneous tissue disorders) | 11 (13) | 16 (18)
arthralgia (Musculoskeletal and connective tissue disorders) | 28 (38) | 45 (66)
myalgia (Musculoskeletal and connective tissue disorders) | 99 (169) | 118 (189)

LIMITATIONS AND CAVEATS:
None reported

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days